CLINICAL TRIAL: NCT05696444
Title: A Prospective, Multi-center, Single-arm Study of the Medtronic Hugo™ Robotic Assisted Surgery (RAS) System in Urologic Surgery (Expand URO)
Brief Title: Medtronic Hugo™ Robotic Assisted Surgery (RAS) System in Urologic Surgery (Expand URO)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDT19051EINURO
Record Dates: First submitted 2022-11-18; First posted 2023-01-25 (Actual); Results first posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Bladder Cancer; Prostate Cancer; Kidney Cancer; Pelvic Tumor; Interstitial Cystitis; Congenital Abnormalities; End Stage Renal Disease; Renal Tumor; Kidney Injury
MeSH Terms: conditions — Urinary Bladder Neoplasms; Prostatic Neoplasms; Kidney Neoplasms; Pelvic Neoplasms; Cystitis, Interstitial; Congenital Abnormalities; Kidney Failure, Chronic; Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Robotic Assisted Surgery (RAS) Urologic Surgery (Other): Robotic Assisted Surgery (RAS) urologic surgery under the umbrella of procedures outlined by the FDA (prostatectomy, cystectomy and nephrectomy).
  Interventions: Device: RAS Prostatectomy; Device: RAS Cystectomy; Device: RAS Nephrectomy

INTERVENTIONS:
Device: RAS Prostatectomy — Subjects indicated for Robotic Assisted Surgery (RAS) for prostatectomy will have RAS surgery using the Medtronic Hugo RAS system.
Device: RAS Cystectomy — Subjects indicated for Robotic Assisted Surgery (RAS) for cystectomy will have RAS surgery using the Medtronic Hugo RAS system.
Device: RAS Nephrectomy — Subjects indicated for Robotic Assisted Surgery (RAS) for nephrectomy (Radical/Partial) will have RAS surgery using the Medtronic Hugo RAS system.

SUMMARY:
This study will evaluate the safety and performance of the Medtronic Hugo™ RAS System when used for urologic RAS procedures.

DETAILED DESCRIPTION:
A prospective, multicenter, single-arm pivotal study in subjects undergoing a urologic RAS procedure using the Medtronic Hugo™ RAS System. Subjects without an oncologic indication will be followed for 30 days post-procedure. Oncologic subjects will be followed annually through 5 years. The study will be conducted in up to 6 investigative sites in the United States of America (USA).

ELIGIBILITY:
Inclusion Criteria:

1. Adult subjects (age ≥ 22 years) as required by local law
2. Subject has been indicated for a radical prostatectomy, radical cystectomy, or nephrectomy (partial or radical) surgical procedure
3. Subject is an acceptable candidate for a fully robotic assisted surgical procedure, a laparoscopic surgical procedure, or an open surgical procedure
4. The subject is willing to participate and consents to participate, as documented by a signed and dated informed consent form

Exclusion Criteria:

1. Subjects for which minimally invasive surgery is contraindicated as determined by the Investigator
2. Subjects with comorbidities or medical characteristics, which would preclude the surgical procedure in the opinion of the Investigator
3. Subjects diagnosed with a bleeding disorder and/or cannot be removed from their anticoagulants prior to surgery based on surgeon discretion and standard-of-care
4. Non-oncology subjects with an estimated life expectancy of less than 6 months; oncology subjects considered for cystectomy with a life expectancy less than 24 months; oncology subjects considered for nephrectomy with a life expectancy less than 60 months; oncology subjects considered for prostatectomy with less than a 10-year life expectancy.
5. Female subjects pregnant at the time of the surgical procedure.
6. Subjects who are considered to be part of a vulnerable population (e.g., prisoners or those without sufficient mental capacity)
7. Subjects who have participated in an investigational drug or device research study within 30 days of enrollment that would interfere with this study
8. Subjects with active infections including but not limited to pneumonia, urinary tract, cellulitis, or bacteremia

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2022-12-14 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2030-01-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Abern, MD, Study Chair — Duke Medical Center
Locations (6):
- United States (6):
  - City of Hope, Duarte, California
  - University of Chiago, Chicago, Illinois
  - Mount Sinai, New York, New York
  - Duke Medical Center, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Swedish Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There was no minimum enrollment requirement at each site; individual sites were not allowed to enroll more than 30% of the total study population. 137 subjects from 6 US sites contributed to the study cohort.
Pre-assignment Details: A total of 144 subjects were consented for enrollment. 7 subjects were discontinued from the study prior to their procedure.
Groups:
- Robotic Assisted Surgery (RAS) Urologic Surgery - Prostatectomy: RAS Prostatectomy: Subjects indicated for Robotic Assisted Surgery (RAS) for prostatectomy will have RAS surgery using the Medtronic Hugo RAS system.
- Robotic Assisted Surgery (RAS) Urologic Surgery - Cystectomy: RAS Cystectomy: Subjects indicated for Robotic Assisted Surgery (RAS) for cystectomy will have RAS surgery using the Medtronic Hugo RAS system.
- Robotic Assisted Surgery (RAS) Urologic Surgery - Nephrectomy: RAS Nephrectomy: Subjects indicated for Robotic Assisted Surgery (RAS) for nephrectomy (Radical/Partial) will have RAS surgery using the Medtronic Hugo RAS system.
Period: Treatment
Arm/Group | Robotic Assisted Surgery (RAS) Urologic Surgery - Prostatectomy | Robotic Assisted Surgery (RAS) Urologic Surgery - Cystectomy | Robotic Assisted Surgery (RAS) Urologic Surgery - Nephrectomy
Started | 55 | 29 | 53
Completed | 55 | 28 | 53
Not Completed | 0 | 1 | 0
Not completed — Physician Decision | 0 | 1 | 0
Period: 30 Days
Arm/Group | Robotic Assisted Surgery (RAS) Urologic Surgery - Prostatectomy | Robotic Assisted Surgery (RAS) Urologic Surgery - Cystectomy | Robotic Assisted Surgery (RAS) Urologic Surgery - Nephrectomy
Started | 55 | 28 | 53
Completed | 53 | 26 | 52
Not Completed | 2 | 2 | 1
Not completed — Death | 1 | 1 | 0
Not completed — Missed Visit | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Robotic Assisted Surgery (RAS) Urologic Surgery - Prostatectomy | Robotic Assisted Surgery (RAS) Urologic Surgery - Cystectomy | Robotic Assisted Surgery (RAS) Urologic Surgery - Nephrectomy | Total
Number analyzed (Participants) | 55 | 29 | 53 | 137
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 33 | 9 | 30 | 72
  >=65 years | 22 | 20 | 23 | 65
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.9 (6.70) | 68.9 (9.24) | 61.2 (10.32) | 63.5 (9.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 20 | 23
  Male | 55 | 26 | 33 | 114
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 2 | 8
  Not Hispanic or Latino | 44 | 19 | 36 | 99
  Unknown or Not Reported | 7 | 8 | 15 | 30
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race, Ethnicity: White | 42 | 20 | 31 | 93
  Race, Ethnicity: Black or African American | 7 | 4 | 14 | 25
  Race, Ethnicity: Asian | 1 | 2 | 5 | 8
  Race, Ethnicity: American Indian or Alaska Native | 0 | 0 | 1 | 1
  Race, Ethnicity: Other | 2 | 1 | 0 | 3
  Race, Ethnicity: Unknown | 3 | 2 | 1 | 6
  Race, Ethnicity: Not Reported | 0 | 0 | 1 | 1
  Race, Ethnicity: Native American or Other Pacific Islander | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: Participants]
  United States | 55 | 29 | 53 | 137

OUTCOME MEASURES:

1. Primary Outcome: Primary Effectiveness Endpoint - Surgical Success Rate, Defined as the Procedure Not Going Into Conversion
Description: The primary effectiveness endpoint is the surgical success rate, defined as the procedure not going into conversion. Conversion is defined as the switch from a robotic assisted approach using the Hugo system to a robotic assisted approach utilizing an FDA cleared robotic-assisted device, laparoscopic, or open surgery.
Time Frame: During surgical procedure
Population: One subject in the cystectomy cohort who met the criteria to be included in the Full Analysis set (FAS), as they received their first incision with intent of using Hugo, was excluded from the analysis as their procedure was aborted after an hour of exploration due to an advanced disease state. Data from the three RAS Urologic Surgery cohorts: Prostatectomy, Cystectomy, & Nephrectomy were combined for analysis per pre-specified analysis plan.
Measure: Count of Participants; unit: Participants
Arm/Group | Robotic Assisted Surgery (RAS) Urologic Surgery
Number analyzed (Participants) | 136
Participants | 134
Statistical Analysis 1: Comparison: Robotic Assisted Surgery (RAS) Urologic Surgery; Test type: Superiority — Test was calculated using an exact test against a null value of 0.85; p < 0.0001, Exact test

2. Primary Outcome: Primary Safety Endpoint - Rate of Subjects With Complications Meeting Grade III - Grade V Criteria Per the Clavien-Dindo Classification System.
Description: Complications meeting Grade III criteria or higher per the Clavien-Dindo Classification system, from first incision through 30 days post-procedure.
  Clavien-Dindo Classification of Surgical Complications:
  Grade I: Any deviation from the normal postoperative course without the need for pharmacological treatment or surgical, endoscopic, and radiological interventions.
  Grade II: Requiring pharmacological treatment with drugs other than such allowed for grade I complications. Blood transfusions and total parenteral nutrition are also included.
  Grade III: Requiring surgical, endoscopic or radiological intervention Grade IIIa: Intervention not under general anesthesia Grade IIIb: Intervention under general anesthesia Grade IV: Life-threatening complication requiring IC/ICU management Grade IVa: Single organ dysfunction (including dialysis) Grade IVb: Multiorgan dysfunction Grade V: Death of a patient
Time Frame: 30 days
Population: Three subjects (1 prostatectomy, 1 cystectomy, 1 nephrectomy) had a missed 30-day follow-up visit.
  Subjects must have met one of the following conditions to be included:
  * They experienced a documented major complication within 30 days of the index procedure, regardless of whether the 30-day visit occurred. OR
  * They completed their 30-day visit, confirming that no major complication occurred.
Measure: Count of Participants; unit: Participants
Arm/Group | Robotic Assisted Surgery (RAS) Urologic Surgery - Prostatectomy | Robotic Assisted Surgery (RAS) Urologic Surgery - Cystectomy | Robotic Assisted Surgery (RAS) Urologic Surgery - Nephrectomy
Number analyzed (Participants) | 54 | 28 | 52
Participants | 2 | 5 | 1
Statistical Analysis 1: Comparison: Robotic Assisted Surgery (RAS) Urologic Surgery - Prostatectomy; Test type: Superiority — Test was calculated using an exact test against a null value of 0.2; p = 0.0006, Exact test — Holm adjusted at alpha = 0.025
Statistical Analysis 2: Comparison: Robotic Assisted Surgery (RAS) Urologic Surgery - Cystectomy; Test was calculated using an exact test against a null value of 0.45; Test type: Superiority; p = 0.0025, Exact test — Holm adjusted at alpha = 0.025
Statistical Analysis 3: Comparison: Robotic Assisted Surgery (RAS) Urologic Surgery - Nephrectomy; Test was calculated using an exact test against a null value of 0.2; Test type: Superiority; p = 0.0001, Exact test — Holm adjusted at alpha = 0.025

3. Secondary Outcome: Secondary Endpoint - Overall Complication Rate From First Incision Through 30 Days Post-procedure.
Description: Complication rate: Overall rate of subjects with one or more complications (Clavien-Dindo Grade I or higher), from the first incision through 30 days post-procedure.
Time Frame: 30 days
Population: Subjects must have met one of the following conditions to be included:
  * They experienced any complication within 30 days of the index procedure, regardless of whether the 30-day visit occurred. OR
  * They completed their 30-day visit, confirming that no complications occurred.
Measure: Count of Participants; unit: Participants
Groups:
- Full Analysis Set (FAS) With Available Data: RAS Prostatectomy: Subjects indicated for Robotic Assisted Surgery (RAS) for prostatectomy will have RAS surgery using the Medtronic Hugo RAS system.
Arm/Group | Full Analysis Set (FAS) With Available Data | Robotic Assisted Surgery (RAS) Urologic Surgery - Cystectomy | Robotic Assisted Surgery (RAS) Urologic Surgery - Nephrectomy
Number analyzed (Participants) | 55 | 29 | 52
Participants | 31 | 24 | 24

4. Secondary Outcome: Secondary Endpoint - Operative Time (Min)
Description: Operative time shall be collected through the length of the procedure.
Time Frame: up to 720 minutes
Population: Operative time, an efficacy measure, is reported only for subjects whose procedures were completed as planned using the Hugo system. This measure excludes aborted cases (n=1 cystectomy) and converted cases (n=2 nephrectomies).
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Robotic Assisted Surgery (RAS) Urologic Surgery - Prostatectomy | Robotic Assisted Surgery (RAS) Urologic Surgery - Cystectomy | Robotic Assisted Surgery (RAS) Urologic Surgery - Nephrectomy
Number analyzed (Participants) | 55 | 28 | 51
Minutes | 227.8 (54.01) | 357.8 (83.26) | 178.7 (69.52)

5. Secondary Outcome: Secondary Endpoint - Intraoperative Estimated Blood Loss (mL).
Description: Intraoperative estimated blood loss shall be collected through the length of the procedure.
Time Frame: intraoperative
Population: Intraoperative Estimated Blood loss, as a safety measure, is reported for all subjects in whom Hugo was utilized during the procedure.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Robotic Assisted Surgery (RAS) Urologic Surgery - Prostatectomy | Robotic Assisted Surgery (RAS) Urologic Surgery - Cystectomy | Robotic Assisted Surgery (RAS) Urologic Surgery - Nephrectomy
Number analyzed (Participants) | 55 | 29 | 53
mL | 161.5 (89.34) | 394.7 (380.29) | 117.5 (122.45)

6. Secondary Outcome: Secondary Endpoint - Transfusion Rate Through 30 Days.
Description: Transfusion rate shall be collected through 30 days post-procedure
Time Frame: 30 days
Population: Transfusion rate, as a safety measure, is reported for all subjects in whom Hugo was utilized during the procedure.
Measure: Count of Participants; unit: Participants
Arm/Group | Robotic Assisted Surgery (RAS) Urologic Surgery - Prostatectomy | Robotic Assisted Surgery (RAS) Urologic Surgery - Cystectomy | Robotic Assisted Surgery (RAS) Urologic Surgery - Nephrectomy
Number analyzed (Participants) | 55 | 29 | 53
Participants | 0 | 9 | 1

7. Secondary Outcome: Secondary Endpoint - Rate of Device-related Conversions
Description: Rate of device-related conversions shall be collected through the length of the procedure.
Time Frame: intraoperative
Population: Rate of Device Related Conversions is reported for all subjects in whom Hugo was utilized during the procedure.
Measure: Count of Participants; unit: Participants
Arm/Group | Robotic Assisted Surgery (RAS) Urologic Surgery - Prostatectomy | Robotic Assisted Surgery (RAS) Urologic Surgery - Cystectomy | Robotic Assisted Surgery (RAS) Urologic Surgery - Nephrectomy
Number analyzed (Participants) | 55 | 29 | 53
Participants | 0 | 0 | 1

8. Secondary Outcome: Secondary Endpoint - Hospital Length of Stay (Days)
Description: Hospital length of stay (days) shall be collected through 30 days post-procedure.
Time Frame: 30 days
Population: Hospital Length of Stay is reported for all subjects in whom Hugo was utilized during the procedure.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Robotic Assisted Surgery (RAS) Urologic Surgery - Prostatectomy | Robotic Assisted Surgery (RAS) Urologic Surgery - Cystectomy | Robotic Assisted Surgery (RAS) Urologic Surgery - Nephrectomy
Number analyzed (Participants) | 55 | 29 | 53
Days | 1.2 (0.9) | 8.4 (11.44) | 1.7 (1.53)

9. Secondary Outcome: Secondary Endpoint - Readmission Rate (Through 30 Days)
Description: Readmission rate shall be collected though 30 days post-procedure.
Time Frame: 30 days
Population: Readmission rate, as a safety measure, is reported for all subjects in whom Hugo was utilized during the procedure.
Measure: Count of Participants; unit: Participants
Arm/Group | Robotic Assisted Surgery (RAS) Urologic Surgery - Prostatectomy | Robotic Assisted Surgery (RAS) Urologic Surgery - Cystectomy | Robotic Assisted Surgery (RAS) Urologic Surgery - Nephrectomy
Number analyzed (Participants) | 55 | 29 | 53
Participants | 2 | 6 | 4

10. Secondary Outcome: Secondary Endpoint - Reoperation Rate (Through 30 Days).
Description: Reoperation rate shall be collected through 30 days post-procedure.
Time Frame: 30 days
Population: Reoperation rate, as a safety measure, is reported for all subjects in whom Hugo was utilized during the procedure.
Measure: Count of Participants; unit: Participants
Arm/Group | Robotic Assisted Surgery (RAS) Urologic Surgery - Prostatectomy | Robotic Assisted Surgery (RAS) Urologic Surgery - Cystectomy | Robotic Assisted Surgery (RAS) Urologic Surgery - Nephrectomy
Number analyzed (Participants) | 55 | 29 | 53
Participants | 0 | 3 | 1

11. Secondary Outcome: Secondary Endpoint - Mortality Rate (Through 30 Days).
Description: Mortality rate shall be collected through 30 days post-procedure.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Robotic Assisted Surgery (RAS) Urologic Surgery - Prostatectomy | Robotic Assisted Surgery (RAS) Urologic Surgery - Cystectomy | Robotic Assisted Surgery (RAS) Urologic Surgery - Nephrectomy
Number analyzed (Participants) | 55 | 29 | 53
Participants | 1 | 1 | 0

12. Secondary Outcome: Secondary Endpoint - Progression-free Survival
Description: Progression-free survival rate will be assessed through 5 years in oncologic subjects.
Time Frame: 5 years
Reporting Status: Not Posted, anticipated posting 2030-01

13. Secondary Outcome: Secondary Endpoint - Disease-free Survival
Description: Disease-free survival rate will be assessed through 5 years in oncologic subjects.
Time Frame: 5 years
Reporting Status: Not Posted, anticipated posting 2030-01

14. Secondary Outcome: Secondary Endpoint - Overall Survival
Description: Overall survival rate will be assessed through 5 years in oncologic subjects.
Time Frame: 5 years
Reporting Status: Not Posted, anticipated posting 2030-01

ADVERSE EVENTS:
Time Frame: All Adverse Events were collected from the time of consent through 30 days post procedure.
Description: All participant deaths within the database snapshot were included.
Groups:
- Robotic Assisted Surgery (RAS) Urologic Surgery - Prostatectomy: RAS Prostatectomy: Subjects indicated for Robotic Assisted Surgery (RAS) for prostatectomy will have the RAS surgery using the Medtronic Hugo RAS system.
- Robotic Assisted Surgery (RAS) Urologic Surgery - Cystectomy: RAS Cystectomy: Subjects indicated for Robotic Assisted Surgery (RAS) for cystectomy will have the RAS surgery using the Medtronic Hugo RAS system.
Arm/Group | Robotic Assisted Surgery (RAS) Urologic Surgery - Prostatectomy | Robotic Assisted Surgery (RAS) Urologic Surgery - Cystectomy | Robotic Assisted Surgery (RAS) Urologic Surgery - Nephrectomy
All-Cause Mortality (participants affected / at risk) | 1/55 | 1/29 | 0/53
Serious Adverse Events (participants affected / at risk) | 5/55 | 15/29 | 7/53
Other Adverse Events (participants affected / at risk) | 19/55 | 7/29 | 6/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Robotic Assisted Surgery (RAS) Urologic Surgery - Prostatectomy (N=55) | Robotic Assisted Surgery (RAS) Urologic Surgery - Cystectomy (N=29) | Robotic Assisted Surgery (RAS) Urologic Surgery - Nephrectomy (N=53)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 7 (7) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Abdominal Hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intestinal Perforation (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0) | 0 (0)
Oedema Peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Anaemia Postoperative (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Arterial Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Incision Site Haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Post Procedural Haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Post Procedural Urine Leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Procedural Haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Wound Dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Post Procedural Hameorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 4 (4) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Urinary Incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Umbilical Haematoma (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 0 | 1 (1) | 0
Lymphocele (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Robotic Assisted Surgery (RAS) Urologic Surgery - Prostatectomy (N=55) | Robotic Assisted Surgery (RAS) Urologic Surgery - Cystectomy (N=29) | Robotic Assisted Surgery (RAS) Urologic Surgery - Nephrectomy (N=53)
Abdominal Pain (Gastrointestinal disorders) | 3 (3) | 2 (2) | 4 (4)
Constipation (Gastrointestinal disorders) | 1 (1) | 3 (3) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 1 (1)
Urinary Incontinence (Renal and urinary disorders) | 16 (16) | 1 (1) | 0 (0)
Erectile Dysfunction (Reproductive system and breast disorders) | 6 (6) | 0/26 (0) | 0/33 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2024-08-21): https://cdn.clinicaltrials.gov/large-docs/44/NCT05696444/Prot_000.pdf
  • Statistical Analysis Plan (2024-11-04): https://cdn.clinicaltrials.gov/large-docs/44/NCT05696444/SAP_001.pdf